CLINICAL TRIAL: NCT03256370
Title: The Association Between Human Milk Oligosaccharide and Development of Allergic Manifestations in Infants
Brief Title: Association of HMOs and Allergic Manifestations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Other Study IDs: HMOs
Record Dates: First submitted 2017-08-11; First posted 2017-08-22 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-04

CONDITIONS: Human Milk Oligosaccharides, Allergic Manifestation
Keywords: Allergic manifestation, Human milk oligosaccharides, Breast Milk

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — human breast-milk

GROUPS / COHORTS (3):
- Infants with allergic diseases: allergic disease : atopic dermatitis or food allergy
  Interventions: Procedure: milk collection
- Healthy infants with atopic mothers: atopic mothers : mothers with asthma or allergic rhinitis or allergic dermatitis (diagnosed by doctors)
  Interventions: Procedure: milk collection
- Healthy infants with non-atopic mothers.: non-atopic mothers : mothers without history of asthma or allergic rhinitis or allergic dermatitis
  Interventions: Procedure: milk collection

INTERVENTIONS:
Procedure: milk collection — * Parents of breast-fed infant from general pediatric clinic and allergy clinic of King Chulalongkorn Memorial Hospital were approached for informed about the research and ask to join this project
  * After completed informed consent, demographic data was collected and filled in case record form
  * Milk of mother in both allergic and control groups were collected 60 ml then transferred to freeze at -80oc to for human milk oligosaccharide analysis
  Method of human milk oligosaccharide analysis :
  1. Ultra High Pressure Liquid Chromatography(UHPLC) with fluorescence method
  2. High-Performance Anion-Exchange Chromatography with Pulsed Amperometric Detection (HPAEC-PAD) method

SUMMARY:
Compare the HMO composition in breast milk of infants with allergic manifestation (atopic dermatitis and food allergy) in the first 3 years of life, healthy infants with allergic mother and healthy infants with non-allergic mother.

DETAILED DESCRIPTION:
* Parents of breast-fed infant from general pediatric clinic and allergy clinic of King Chulalongkorn Memorial Hospital were approached for informed about the research and ask to join this project
* After completed informed consent, demographic data was collected and filled in case record form
* Milk of mother in both allergic and control groups were collected 60 ml then transferred to freeze at -80oc to for human milk oligosaccharide analysis

ELIGIBILITY:
Inclusion Criteria:

1. mothers with breast-fed infant with or without allergic manifestation
2. Intend to participate for follow up and sign consent to participate in the study

Exclusion Criteria:

1. Mothers with any medical illness or high risk infant pregnant
2. Infants with disease which affected allergic disease
3. No inform consent
4. Anything in the opinion of the investigator that would prevent children from completing the study

Max Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Normal term children (born after 37 weeks gestation) from low risk healthy pregnant women aged 18-40 years divided to 3 groups i. Allergic groups : infants with allergic manifestation ii. High risk control groups : atopic mother with infant no disease iii. Healthy control groups : non- atopic mother with infant no disease
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-10-05 (Estimated); Study Completion 2019-10-05 (Estimated)

PRIMARY OUTCOMES:
Atopic dermatitis | first 2 years of life
  Relapsing eczematous typical morphology on typical distribution (Scalp, face, neck, and extensor surfaces of the skin) Typical morphology Acute and subacute : erythematous papules and plaques, may vesiculate and become exudative Chronic : lichenification, papules and excoriations
IgE mediated food allergy | first 2 years of life
  confirmed by oral food challenge
Non-IgE mediated food allergy | first 2 years of life
  Presentation of clinical ex. bloody stool when repeating episode occurred with the same food more than twice. Improvement of symptom after eliminating of suspected food

CONTACTS AND LOCATIONS:
Locations (1):
- Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided